CLINICAL TRIAL: NCT00900172
Title: Angiogenesis Pathway Gene Polymorphisms Associated With Clinical Outcome in Patients Enrolled in ECOG 4599
Brief Title: Study of Blood and Tissue Samples From Patients With Locally Advanced, Metastatic, or Recurrent Non-Small Cell Lung Cancer Treated With Bevacizumab, Carboplatin, and Paclitaxel
Status: Completed | Type: Observational
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Other Study IDs: CDR0000592945; ECOG-E4599T1
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer; adenocarcinoma of the lung; bronchoalveolar cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Bevacizumab; Carboplatin; Paclitaxel; Gene Expression Profiling; Polymerase Chain Reaction; Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Biological: bevacizumab
Drug: carboplatin
Drug: paclitaxel
Genetic: gene expression analysis
Genetic: polymerase chain reaction
Genetic: polymorphism analysis
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood and tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This research study is looking at blood and tissue samples from patients with locally advanced, metastatic, or recurrent non-small cell lung cancer treated with bevacizumab, carboplatin, and paclitaxel.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine whether germline polymorphisms (DNA) of genes involved in DNA repair (e.g., XPD, ERCC-1, and others) and angiogenesis (e.g., vascular endothelial growth factor [VEGF], interleukin-8, CXCR2, adrenomedullin, leptin, and others) are associated with toxicity and clinical outcome in patients with non-small cell lung cancer enrolled on protocol ECOG-4599.

OUTLINE: Blood samples previously obtained from patients on protocol ECOG-4599 are analyzed for the association of germline variations of genes involved in DNA repair (XPD and ERCC1), angiogenesis (VEGF and IL-8), and clinical outcome (overall survival, response, progression-free survival, and toxicity).

Tumor cells are collected from paraffin-embedded tissue using laser-capture microdissection and normal tissue is collected from the specimen. Polymorphisms in ERCC-1, XRCC-1, XRCC-3, GST-P1, TGF-β, and IL-8CXCR are assessed using Taqman assays.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Available serum or plasma samples from patients with locally advanced, metastatic, or recurrent non-squamous non-small cell lung cancer

  * Stage IIIB (with pleural effusion) or stage IV disease
* Enrolled on protocol ECOG-4599

  * Treated with carboplatin and paclitaxel with or without bevacizumab

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples submitted for research from patients participating in E4599
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2008-03-15 (Actual); Primary Completion 2009-04-15 (Actual); Study Completion 2009-04-15 (Actual)

PRIMARY OUTCOMES:
Correlation of results to response and toxicity | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Heinz-Josef Lenz, MD, Study Chair — University of Southern California